CLINICAL TRIAL: NCT03772522
Title: The Identity Project: An Evaluation of an Identity Capital Intervention for Young People Transitioning Out of Homelessness
Brief Title: The Identity Project
Acronym: TIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: dk Leadership (Industry); Covenant House Toronto (Other); Ontario Trillium Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-002
Record Dates: First submitted 2018-09-23; First posted 2018-12-11 (Actual); Results first posted 2020-05-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Youth; Homelessness
Keywords: Hopelessness; Self Esteem; Social Isolation; Employment Status; Education; Housing Problems; Identity, Social; Self Efficacy; Control Locus; Poverty; Youth; Homelessness; Homeless Youth
MeSH Terms: conditions — Social Isolation; Social Identification

STUDY DESIGN:
Intervention Model Description: Thirty young people (aged 18 - 26 years) who have transitioned out of homelessness within the past three years will be offered scholarships to participate in a six-week intervention that focuses on building identity capital and providing career direction. The intervention will be designed and carried out by dk Leadership - an established, highly successful leadership and counseling centre in Toronto with a track record of significantly improving the life trajectories of teens and adults. Importantly, study participants will be incorporated into the centre's current programming, meaning the intervention will be held at a location not associated with homelessness. All of the participants will be invited to attend two focus groups, which will be conducted immediately post-intervention and at six months post-intervention. Each focus group will contain approximately 8 - 10 youth. Participants in the intervention and delayed intervention will be in separate focus groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate dk Leadership Intervention (Experimental): Participants allocated to the immediate intervention group are assessed for study outcomes immediately prior to the 6-week dk Leadership intervention and immediately after the intervention.
  Outcomes measured immediately post-intervention are compared with participants who have not received the intervention during the 6 weeks.
  After the delayed intervention group takes the intervention, the two groups are joined into a single arm.
  Interventions: Behavioral: dk Leadership
- Delayed dk Leadership Intervention (Placebo Comparator): Participants allocated to this arm receive 6 weeks of no intervention. Outcomes are measured immediately before and immediately after the 6 week period. The change in outcomes are compared with participants who have received the intervention during the 6 week period.
  This group then receives the same dk Leadership intervention; after this point, the two groups are joined into a single arm for subsequent analyses.
  Interventions: Behavioral: dk Leadership

INTERVENTIONS:
Behavioral: dk Leadership — Participants will attend two full-day workshops and four half-day group coaching sessions over the course of six weeks. The workshops and coaching sessions will be supplemented by on-line (e.g., podcasts) and print (e.g., workbooks) material. The full-day workshops will focus on identity-enhancing topics such as self-understanding, creating a life of meaning and purpose, and strategic career development. The half-day group coaching sessions will focus on workshop debriefing and on exploring solutions to transition-related challenges faced by study participants. The program was designed and carried out by dk Leadership - an established leadership and executive coaching centre in Toronto, Canada.

SUMMARY:
Understanding how to create successful pathways out of homelessness is crucial. Thirty young people (aged 18 - 26 years) who have transitioned out of homelessness within the past three years will be offered scholarships to participate in a six week intervention that focuses on building identity capital (sense of purpose and control, self-efficacy and self-esteem) and providing career direction. The intervention will be designed and carried out by dk Leadership - an established, highly successful leadership and counseling centre in Toronto with a track record of significantly improving the life trajectories of teens and adults. Importantly, study participants will be incorporated into the centre's current programming, meaning the intervention will be held at a location not associated with homelessness. Study participants will be collaboratively recruited by dk Leadership and Covenant House Toronto - Canada's largest agency for street-involved and homeless youth.

This impact and process evaluation aims to address critical gaps in knowledge about transition-related supports by asking whether and how an identity capital intervention delivered outside the social service sector impacts the life-trajectories of formerly homeless young people. Particular attention will be paid to whether this intervention shows promise as an unconventional way to tackle poverty and improve social inclusion.

It is hypothesize that, for the primary quantitative outcome measures of hope, community integration, social connectedness, and self-esteem:

1. Significant improvements in the mean scores of the intervention group compared to the delayed intervention comparison group immediately post-intervention will be observed.
2. Significant improvements in the mean scores of both groups (intervention and delayed intervention) immediately post-intervention will be observed.
3. These significant improvements will be sustained in both groups for at least three months post-intervention.

DETAILED DESCRIPTION:
Young people comprise almost 20% of the homeless population in Canada. It is estimated between 35,000 and 40,000 Canadian youth (aged 13 - 25 years) are homeless at some point during the year and at least 6,000 on any given night. In Toronto, an estimated 1,000 - 2,000 youth find themselves searching for a place to sleep on any given night.

While a great deal is known about the risk factors associated with young people entering and remaining entrenched in street life (e.g., intergenerational poverty, childhood abuse, inadequate education, and limited employment opportunities), less is known much less about how to facilitate and sustain transitions off the streets for youth experiencing homelessness.

The scarcity of evidence on this issue means there are critical gaps in understanding how best to help homeless young people move forward in life after they become housed. For example, results from a recent longitudinal mixed method study of 51 formerly homeless youth living in Toronto and Halifax - led by Dr. Sean Kidd and colleagues and one of the most rigorous investigations to date - showed that obtaining stable housing did not necessarily translate into a sense of belonging or connection to mainstream society. While study participants demonstrated incredible commitment, the structural barriers they experienced during the transition process (e.g., inadequate education and underemployment) led to fragile identities (i.e., self-concept) as they experienced a significant decline in hope and a sense of being 'stuck'. Youth described feeling unprepared for and overwhelmed by the realities associated with the transition process, undermining their sense of belonging and confidence in achieving larger life goals.

Building on the Kidd et al. study, Dr. Naomi Thulien (the lead investigator for this study) spent 10 months following nine young people who had left the shelter system and moved into market rent housing in Toronto. The study - believed to be the first of its kind - captured the crucial role identity plays in the transition away from homelessness. Despite their remarkable determination, study participants lacked sufficient identity capital - conceptualized as a sense of purpose and control, self-efficacy, and self-esteem - to help them press on in the face of significant structural inequities. Thulien asserts that failure to understand and incorporate identity capital into transition-related supports may result in a poor return on investment as these supports are likely to be ineffective, underutilized, or rejected outright.

One notable identity-based intervention is a randomized controlled trial that targeted 264 eighth graders from high-poverty and high-unemployment neighborhoods in Detroit, Michigan. Participants who attended the seven-week intervention aimed at aligning the students' current identities with achievable positive adult identities, demonstrated improved outcomes on measures pertaining to academics, mood, and behavior, which was sustained through the two-year follow-up. The authors suggest brief identity-based interventions can have significant effects on outcomes. Despite being suggested as a promising approach, the investigators know of no other interventions (nationally or internationally) that are specifically targeting the enhancement of identity capital for formerly homeless young people. Given the limited evidence-based interventions for youth transitioning out of homelessness, the investigators believe there is a critical need for evaluations that compare findings based on different approaches, reflecting the diversity of the population and their corresponding needs.

The proposed intervention is based on two premises: 1) identity is socially constructed and malleable; and 2) people act in identity-congruent ways. Thus, the intervention aims to change socially constructed life trajectories by providing identity-enhancing resources to formerly homeless young people.

This impact and process evaluation aims to address critical gaps in the literature about transition-related supports by asking whether and how an identity capital intervention delivered outside the social service sector impacts the life-trajectories of formerly homeless young people. Particular attention will be paid to whether this intervention shows promise as an unconventional way to tackle poverty and improve social inclusion.

Specifically, this evaluation will investigate and disseminate important new knowledge on the following outcomes

1. The impact of the intervention on measures of hope, community integration, social connectedness, and self-esteem.
2. The effectiveness of the intervention to increase the number of young people in education, employment, or training.
3. Understanding any practical challenges encountered during the intervention implementation and how these challenges were resolved.
4. Understanding what young people found most beneficial about the intervention and their suggestions for how it could be improved.

An impact and process evaluation utilizing a mixed method prospective cohort design with an intervention and delayed intervention comparison group is the most appropriate because it:

1. Addresses the crucial need to understand and disseminate evidence regarding the impact and process of interventions targeting homeless youth - both will help assess and inform questions related to scalability.
2. Provides a more complete and synergistic utilization of data.
3. Balances scientific rigor with the ethical principle of fairness.

This evaluation is a mixed-methods design with a strong qualitative component. Quantitative data collection will occur at six weeks pre-baseline (for the delayed intervention group only), baseline (immediately pre-intervention), immediately post-intervention (one week), three months post-intervention, six months post-intervention, and nine months post-intervention. At each data collection period, participants will be asked whether they are enrolled in education, employment, or training in the questionnaire. They will also be asked about their housing status. Hope, community integration, social connectedness, and self-esteem will be measured quantitatively using scales.

The frequencies, means and standard deviations will be calculated for all evaluation variables. To address the question about the extent to which the outcome variables change over time, independent t-tests will be conducted on the continuous variables (hope, community integration, social connectedness, and self-esteem) and chi-square tests on the categorical variables (education, employment, training, and housing) to report on changes between: 1) baseline and immediately post-intervention; 2) baseline and three months post-intervention; 3) baseline and six months post-intervention; and 4) baseline and nine months post-intervention. To address the question about whether the intervention group demonstrates a statistically significant difference in outcomes compared to no intervention, the outcome variables between the intervention group and the delayed intervention group will be compared six weeks after the baseline questionnaires (i.e., the intervention group will have just completed the dk Leadership program and the delayed intervention group will not have started it yet).

Qualitative measures are an important feature of this evaluation and will consist of: 1) participant observation and 2) focus groups.

Over the six-week intervention period, the co-investigator will attend the weekly meetings as an observer. She will do this with both the intervention and the delayed intervention group. During these meetings, the investigator will take field notes, documenting her perceptions about the way the workshops and group coaching sessions are being run, and how they are being 'taken up' by the young people in the intervention group.

Focus groups, will take place immediately (one week), three months, six months, and 9 months post-intervention. Participants in the intervention and delayed intervention will be in separate focus groups. The questions posed during the focus groups will be guided by the evaluation objectives, but will be conversational and exploratory in nature with particular attention to identity capital, life-trajectories, and social inclusion. It is anticipated that the focus groups will last 60 - 90 minutes. All will be conducted by the co-investigator at locations most convenient for the study participants, and will be audio recorded and transcribed verbatim.

In keeping with the emergent, iterative nature of research using a qualitative design, data analysis and interpretation will begin at the onset of the intervention. The handwritten field notes from the participant observation sessions will be typed into Microsoft Word by the co-investigator immediately after each biweekly meeting. The focus groups will be audio recorded and transcribed verbatim. In order to conduct a more nuanced analysis of the data, the transcriptionist will be instructed to note short responses, uncooperative tones, and literal silence. Prior to each meeting with the participants, the co-investigator will conduct a preliminary data analysis, reading the field notes multiple times, separating the data into coded segments, making analytic memos beside large portions of the field notes or transcripts, identifying emerging themes (and comparing/contrasting these between participants), and complying new questions to ask the participants. Participants will be asked for their perspectives on the emerging interpretations at each visit and these perspectives will play a key role in helping shape the data analysis and help ensure the trustworthiness of the data. The web-based application Dedoose39 will be utilized to assist with sorting and coding the qualitative data.

Study participants may benefit from the opportunity to share with the co-investigator and with each other about whether and how an identity-building intervention delivered outside the social service sector impacts their life-trajectories. Additionally, participants may derive satisfaction from knowing that their contributions will help advance understanding about how best to design interventions that help tackle poverty and improve social inclusion for young people transitioning out of homelessness.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-26 years of age
* Left homelessness within the last 3 years (youth living in supportive housing contexts (e.g., transitional housing) will be considered to have left homelessness)
* Currently not homeless (youth in supportive or transitional housing are eligible)
* A concerted effort will be made to recruit young people facing additional identity-related challenges like newcomer and racialized youth, Indigenous youth, and youth who belong to the LGBTQ2S community.

Exclusion Criteria:

* Not fluent in English
* Cannot provide informed consent
* Cannot commit to attending two full-day workshops and four half-day group coaching sessions over the course of six weeks (missing more than one workshop and two coaching sessions will disqualify participants from the study)

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-06 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi S Thulien, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaetz, S., Dej, E., Richter, T., & Redman, M. (2016) The state of homelessness in Canada 2016. Toronto, ON: Canadian Observatory on Homelessness Press. Retrieved from http://www.homelesshub.ca/SOHC2016
- [Background] Gaetz, S., & Redman, M. (2016). Federal investment in youth homelessness: Comparing Canada and the United States and a proposal for reinvestment. Canadian observatory on homelessness policy brief. Toronto, ON: The Homeless Hub Press. Retrieved from http://homelesshub.ca/sites/default/files/Policy_Brief.pdf
- [Background] Karabanow, J. (2008). Getting off the street: Exploring the process of young people's street exits. American Behavioral Scientist, 51(6), 772-788. doi:10.1177/0002764207311987
- [Background] Covenant House Toronto. (2016). Facts and stats. Retrieved from http://www.covenanthousetoronto.ca/homeless-youth/Facts-and-Stats
- [Background] Kidd, S.A., Frederick, T., Karabanow, J., Hughes, J., Naylor, T., & Barbic, S. (2016). A mixed methods study of recently homeless youth efforts to sustain housing and stability. Child and Adolescent Social Work Journal, 33(3), 207-218. doi:10.1007/s10560-015-0424-2
- [Background] Mayock, P., O'Sullivan, E., & Corr, M.L. (2011). Young people exiting homelessness: An exploration of process, meaning and definition. Housing Studies, 26(6), 803-826. doi:10.1080/02673037.2011.593131
- [Background] Brueckner, M., Green, M., & Saggers, S. (2011). The trappings of home: Young homeless people's transitions towards independent living. Housing Studies, 26(1), 1-16. doi:10.1080/02673037.2010.512751
- [Background] Thulien NS, Gastaldo D, Hwang SW, McCay E. The elusive goal of social integration: A critical examination of the socio-economic and psychosocial consequences experienced by homeless young people who obtain housing. Can J Public Health. 2018 Feb;109(1):89-98. doi: 10.17269/s41997-018-0029-6. PMID 29981071
- [Background] Altena AM, Brilleslijper-Kater SN, Wolf JL. Effective interventions for homeless youth: a systematic review. Am J Prev Med. 2010 Jun;38(6):637-45. doi: 10.1016/j.amepre.2010.02.017. PMID 20494240
- [Background] Coren E, Hossain R, Pardo JP, Veras MM, Chakraborty K, Harris H, Martin AJ. Interventions for promoting reintegration and reducing harmful behaviour and lifestyles in street-connected children and young people. Evid Based Child Health. 2013 Jul;8(4):1140-272. doi: 10.1002/ebch.1923. PMID 23877940
- [Background] Hwang SW, Burns T. Health interventions for people who are homeless. Lancet. 2014 Oct 25;384(9953):1541-7. doi: 10.1016/S0140-6736(14)61133-8. PMID 25390579
- [Background] Gaetz, S. (2014). Coming of age: Reimagining the response to youth homelessness in Canada. Toronto, ON: The Canadian Homelessness Research Network Press. Retrieved from http://www.homelesshub.ca/comingofage
- [Background] Karabanow, J., Carson, A., & Clement, P. (2010). Leaving the streets: Stories of Canadian youth. Halifax, NS: Fernwood Publishing.
- [Background] Public Interest. (2009). Changing patterns for street involved youth. Toronto, ON: Author. Retrieved from http://www.worldvision.ca/Programs-and- Projects/Canadian Programs/Documents/ChangingPatternsForStreetInvolvedYouth.pdf
- [Background] Milburn NG, Rice E, Rotheram-Borus MJ, Mallett S, Rosenthal D, Batterham P, May SJ, Witkin A, Duan N. Adolescents Exiting Homelessness Over Two Years: The Risk Amplification and Abatement Model. J Res Adolesc. 2009 Dec 1;19(4):762-785. doi: 10.1111/j.1532-7795.2009.00610.x. PMID 25067896
- [Background] Karabanow, J., Kidd, S., Frederick, T., & Hughes, J. (2016). Toward housing stability: Exiting homelessness as an emerging adult. Journal of Sociology & Social Welfare, 43(1), 121- 148. Retrieved from https://wmich.edu/socialworkjournal
- [Background] Frederick, T., Chwalek, M., Hughes, J., Karabanow, J., & Kidd, S. (2014). How stable is stable? Defining and measuring housing stability. Journal of Community Psychology, 42(8), 964- 979. doi:10.1002/jcop.21665
- [Background] Thulien, N.S. (2017). Chronic precarity: A critical examination of homeless youth transitions to independent housing (Doctoral dissertation). University of Toronto: Toronto, ON. Retrieved from https://tspace.library.utoronto.ca/bitstream/1807/78804/3/Thulien_Naomi_201706_PhD_thesis.pdf
- [Background] Côté, J.E. (2016). The identity capital model: A handbook of theory, methods, and findings. Unpublished manuscript, Department of Sociology, The University of Western Ontario, London, Ontario, Canada. Retrieved from https://www.researchgate.net/publication/305698905_The_Identity_Capital_Model_A_Handbook_Of_Theory_Methods_And_Findings
- [Background] Oyserman D, Bybee D, Terry K. Possible selves and academic outcomes: How and when possible selves impel action. J Pers Soc Psychol. 2006 Jul;91(1):188-204. doi: 10.1037/0022-3514.91.1.188. PMID 16834488
- [Background] Lee, C., & Berrick, J.D. (2014). Experiences of youth who transition to adulthood out of care: Developing a theoretical framework. Children and Youth Services Review, 46, 78-84. Retrieved from http://dx.doi.org/10.1016/j.childyouth.2014.08.005
- [Background] Kidd, S., Frederick, T., Morales, S., Daley, M., & Vitopoulos, N. (2016, November). The Toronto housing outreach program collaborative (HOP-C): Stabilizing housing for recently homeless youth. Oral presentation at the Canadian Alliance to End Homelessness National Conference, Montreal, QC. Retrieved from http://conference.caeh.ca/wp-content/uploads/AWH5_The-Toronto-Housing-Outreach-Program-Collaborative-TFrederick-et-al.pdf
- [Background] Oyserman D, Destin M. Identity-based motivation: Implications for intervention. Couns Psychol. 2010 Oct;38(7):1001-1043. doi: 10.1177/0011000010374775. PMID 21516204
- [Background] Cote JE, Schwartz SJ. Comparing psychological and sociological approaches to identity: identity status, identity capital, and the individualization process. J Adolesc. 2002 Dec;25(6):571-86. doi: 10.1006/jado.2002.0511. PMID 12490176
- [Background] dkLeadership. (2017). Dream it. Do it. Retrieved from http://www.dkleadership.org Urbaniak, G.C., & Plous,S. (2013). Research Randomizer (Version 4.0) [Computer software]. Retrieved from https://www.randomizer.org
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Background] Stergiopoulos V, Gozdzik A, O'Campo P, Holtby AR, Jeyaratnam J, Tsemberis S. Housing First: exploring participants' early support needs. BMC Health Serv Res. 2014 Apr 13;14:167. doi: 10.1186/1472-6963-14-167. PMID 24725374
- [Background] Lee, R. M., & Robbins S. B. (1995). Measuring belongingness: The social connectedness and the social assurance scales. Journal of Counseling Psychology, 42, 232-241
- [Background] Rosenberg, M. (1965). Society and the adolescent self-image. Princeton, NJ: Princeton University Press.
- [Background] Hammersley, M., & Atkinson, P. (2007). Ethnography: Principles in Practice (3rd ed.). London, UK: Routledge.
- [Background] Kusenbach, M. (2003). Street phenomenology: The go-along as ethnographic research tool. Ethnography, 4(3), 455-485. Retrieved from http://eth.sagepub.com
- [Background] Creswell, J.W. (2014). Research design: Qualitative, quantitative, and mixed method approaches (4th ed.). Thousand Oaks, CA: Sage.
- [Background] Eakin JM, Mykhalovskiy E. Reframing the evaluation of qualitative health research: reflections on a review of appraisal guidelines in the health sciences. J Eval Clin Pract. 2003 May;9(2):187-94. doi: 10.1046/j.1365-2753.2003.00392.x. PMID 12787182
- [Background] Kawabata, M., & Gastaldo, D. (2015). The less said, the better: Interpreting silence in qualitative research. International Journal of Qualitative Research Methods, 14(4), 1-9. doi:10.1177/1609406915618123
- [Background] Loiselle, C.G., Profetto-McGrath, J., Polit, D.F., & Tatano Beck, C.T. (2004). Canadian essentials of nursing research. Philadelphia, PA: Lippincott Williams & Wilkins.
- [Background] SocioCultural Research Consultants, LLC. (2016). Dedoose (Version 7.0.23) [web application]. Retrieved from http://www.dedoose.com
- [Result] Thulien NS, Wang A, Mathewson C, Wang R, Hwang SW. Tackling exclusion: A pilot mixed method quasi-experimental identity capital intervention for young people exiting homelessness. PLoS One. 2021 Aug 20;16(8):e0256288. doi: 10.1371/journal.pone.0256288. eCollection 2021. PMID 34415951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between March, 2018 and September, 2018. Participants were collaboratively recruited by our community partner Covenant House Toronto, who referred youth to our research team.
Pre-assignment Details: Although out recruitment goal was 26 youth, we exceeded that goal by recruiting 27 youth.
Groups:
- Immediate dk Leadership Intervention: Participants allocated to the immediate intervention group are assessed for study outcomes immediately before and after the intervention.
  Outcomes measured immediately post-intervention are compared with participants who have not received the intervention during the 6 weeks. After the delayed intervention group takes the intervention, the two groups are joined into a single arm.
  dk Leadership: Participants will attend two full-day workshops and four half-day group coaching sessions over the course of six weeks. The full-day workshops will focus on identity-enhancing topics such as self-understanding, creating a life of meaning and purpose, and strategic career development. The half-day group sessions will focus on workshop debriefing and on exploring solutions to transition-related challenges faced by study participants. The program was designed and carried out by dk Leadership - an established leadership and executive coaching centre in Toronto, Canada.
- Delayed dk Leadership Intervention: Participants allocated to this arm receive 6 weeks of no intervention. Outcomes are measured immediately before and after the 6 week period. The change in outcomes are compared with participants who have received the intervention during the 6 week period.
  This group then receives the same dk Leadership intervention; after this point, the two groups are joined into a single arm for subsequent analyses.
  dk Leadership: Participants will attend two full-day workshops and four half-day group coaching sessions over the course of six weeks. The full-day workshops will focus on identity-enhancing topics such as self-understanding, creating a life of meaning and purpose, and strategic career development. The half-day group sessions will focus on workshop debriefing and on exploring solutions to transition-related challenges faced by study participants. The program was designed and carried out by dk Leadership - an established leadership and executive coaching centre in Toronto, Canada.
Period: Pre-intervention
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention
Started | 12 | 15
Completed | 9 | 11
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 3 | 4
Period: Intervention
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention
Started | 9 | 11
Completed | 8 | 11
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Post-intervention Follow-up
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention
Started | 8 | 11
Completed | 7 | 11
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.5 (3.1) | 23.2 (1.3) | 22.9 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 2 | 6 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 4
  Black/African Canadian | 4 | 3 | 7
  Asian (East Asian, South Asian, Middle Eastern) | 1 | 3 | 4
  Other | 1 | 3 | 4
Immigration Status [Count of Participants; unit: Participants]
  Canadian Citizen | 6 | 7 | 13
  Permanent Resident | 1 | 4 | 5
  Refugee | 1 | 0 | 1
Highest Level of Education Obtained [Count of Participants; unit: Participants]
  Less than high school | 2 | 2 | 4
  Completed high school | 2 | 6 | 8
  Some or complete post-secondary | 4 | 3 | 7
Social Assistance [Count of Participants; unit: Participants]
  Not receiving social assistance | 2 | 2 | 4
  Unemployment benefit | 4 | 4 | 8
  Disability benefit | 2 | 5 | 7
Pursuing Education, Employment or Training [Count of Participants; unit: Participants]
  Currently pursuing EET | 7 | 7 | 14
  Not pursuing EET | 1 | 4 | 5
Current Living Situation [Count of Participants; unit: Participants]
  Market housing | 2 | 5 | 7
  Transitional housing | 3 | 1 | 4
  Social or subsidized housing | 2 | 5 | 7
  Living with family | 1 | 0 | 1
Monthly Rent [Count of Participants; unit: Participants]
  $0-$499 | 4 | 7 | 11
  $500-$999 | 4 | 2 | 6
  $1000+ | 0 | 2 | 2
Years Lived Apart from Family [Count of Participants; unit: Participants]
  <4 | 5 | 4 | 9
  >=4 | 3 | 7 | 10
Number of Attempts at Leaving Homelessness [Count of Participants; unit: Participants]
  <2 | 2 | 7 | 9
  >=2 | 6 | 4 | 10
Family Involvement with a Child Protection Agency [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 4
  No | 5 | 10 | 15
Lived in a Foster or Group Home [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 2
  No | 7 | 10 | 17
Has Children [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 2
  No | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hopelessness as Measured by the Beck Hopelessness Scale
Description: Assessed using Beck's Hopelessness Scale, a 20-item scale which measures motivation, expectations, and feelings about the future (internal consistency α = .93). The total scoring range is 0-20, with 0-3 = no or minimal hopelessness, 4-8 = mild hopelessness, 9-14 = moderate hopelessness- requires monitoring, and 15+ = severe hopelessness- suicide risk.
  Participants' scores at baseline will be compared with their scores post-intervention to detect changes in levels of hopelessness. The change in scores over time will describe the general trajectory of hopelessness.
Time Frame: Assessed at 6 weeks pre-baseline (for the delayed intervention group only), at baseline (immediately pre-intervention), immediately post-intervention, 3 months post-intervention, 6 months post-intervention, and 9 months post-intervention
Population: 1 participant in the delayed intervention group missed the 6-week delay period and joined immediately pre-intervention.Thus, the number of participants at 6-weeks pre-baseline is 10 rather than 11.
  1 participant was lost to follow-up at the 9-month follow-up. Thus the number of participants in the immediate intervention group was 7 rather than 8.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Immediate dk Leadership Intervention: Participants receive the dk Leadership intervention immediately after their baseline interview.
  dk Leadership: Participants will attend two full-day workshops and four half-day group coaching sessions over the course of six weeks. The full-day workshops will focus on identity-enhancing topics such as self-understanding, creating a life of meaning and purpose, and strategic career development. The half-day group sessions will focus on workshop debriefing and on exploring solutions to transition-related challenges faced by study participants. The program was designed and carried out by dk Leadership - an established leadership and executive coaching centre in Toronto, Canada.
- Delayed dk Leadership Intervention: Participants allocated to this arm are followed for 6 weeks after enrolment with no intervention; they then receive the dk Leadership intervention.
  dk Leadership: Participants will attend two full-day workshops and four half-day group coaching sessions over the course of six weeks. The full-day workshops will focus on identity-enhancing topics such as self-understanding, creating a life of meaning and purpose, and strategic career development. The half-day group sessions will focus on workshop debriefing and on exploring solutions to transition-related challenges faced by study participants. The program was designed and carried out by dk Leadership - an established leadership and executive coaching centre in Toronto, Canada.
- Pooled Analysis of Immediate and Delayed Intervention Groups: After both groups had received the dk Leadership intervention, analyses for the immediate and delayed intervention groups were pooled for subsequent analyses. These timepoints include immediately post-intervention, 3-months post-intervention, 6-months post-intervention and 9-months post-intervention.
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 8 | 11 | 19
score on a scale
  6-weeks pre-baseline: number analyzed (Participants) | 8 | 10 | 18
  6-weeks pre-baseline | NA (NA) — Data wasn't taken for the immediate intervention group at this timepoint. | 6.70 (4.08) | NA (NA) — Data wasn't taken for the immediate intervention group at this timepoint.
  Baseline (pre-intervention) | 4.27 (3.28) | 6.55 (3.80) | 5.59 (3.68)
  Immediately post-intervention | 2.63 (3.46) | 5.21 (4.01) | 4.12 (3.92)
  3 Months post-intervention | 2.75 (2.71) | 5.55 (3.80) | 4.36 (3.59)
  6 Months post-intervention | 1.75 (1.98) | 5.01 (3.57) | 3.64 (3.37)
  9 Months post-intervention: number analyzed (Participants) | 7 | 11 | 18
  9 Months post-intervention | 1.71 (1.70) | 5.00 (4.20) | 3.72 (3.75)
Statistical Analysis 1: Comparison: Immediate dk Leadership Intervention vs Delayed dk Leadership Intervention; Change in score in the immediate intervention group (after receiving the intervention for 6 weeks) compared to that of the delayed intervention group (after receiving no intervention for 6 weeks); Test type: Superiority; p = 0.428, t-test, 2 sided; Cohen's d (effect size) = 0.384
Statistical Analysis 2: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of scores at baseline (pre-intervention) and immediately post-intervention; Test type: Superiority; p = 0.058, t-test, 2 sided; Cohen's d (effect size) = -0.46
Statistical Analysis 3: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of scores at baseline (pre-intervention) and 3-month post-intervention; Test type: Superiority; p = 0.095, t-test, 2 sided; Cohen's d (effect size) = -0.40
Statistical Analysis 4: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of scores at baseline (pre-intervention) and 6-months post-intervention; Test type: Superiority; p = 0.005, t-test, 2 sided; Cohen's d (effect size) = -0.73
Statistical Analysis 5: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of scores at baseline (pre-intervention) and 9-months post-intervention; Test type: Superiority; p = 0.022, t-test, 2 sided; Cohen's d (effect size) = -0.60

2. Primary Outcome: Mean Change From Baseline in Community Integration (Psychological and Physical) Scores as Measured by the Community Integration Scale (CIS)
Description: Assessed using the Community Integration Scale, an 11-item scale which measures behavioural (e.g., participation in activities) and psychological (e.g., sense of belonging) aspects of community integration. The CIS includes a physical subscale (with scores ranging from 0-7) and a psychological subscale (with scores ranging from 4-20). Higher scores indicate greater community integration. This scale was used extensively in the Chez Soi/At Home study, but psychometric properties have yet to be reported.
  Participants' scores at baseline will be compared with their scores post-intervention to detect changes in levels of community integration. The change in scores over time will describe the general trajectory of community integration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pooled Analysis of Immediate and Delayed Intervention Groups: After both groups had received the dk Leadership intervention, analyses for the immediate and delayed intervention groups were pooled for subsequent analyses. Analyses were performed immediately post-intervention, 3-months post-intervention, 6-months post-intervention and 9-months post-intervention
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 8 | 11 | 19
score on a scale
  Physical sub-scale: 6-weeks pre-baseline: number analyzed (Participants) | 8 | 10 | 18
  Physical sub-scale: 6-weeks pre-baseline | NA (NA) — Data wasn't taken for the immediate intervention group at this timepoint. | 4.42 (2.12) | NA (NA) — Data wasn't taken for the immediate intervention group at this timepoint.
  Physical sub-scale: Baseline (pre-intervention) | 2.50 (1.20) | 3.09 (2.30) | 2.84 (1.89)
  Physical sub-scale: Immediately post-intervention | 3.89 (1.11) | 3.45 (1.86) | 3.64 (1.57)
  Physical sub-scale: 3 Months post-intervention | 3.98 (2.37) | 3.55 (2.07) | 3.73 (2.14)
  Physical sub-scale: 6 Months post-intervention | 3.75 (1.91) | 3.64 (1.50) | 3.68 (1.63)
  Physical sub-scale: 9 Months post-intervention: number analyzed (Participants) | 7 | 11 | 18
  Physical sub-scale: 9 Months post-intervention | 3.29 (2.36) | 3.45 (1.57) | 3.39 (1.85)
  Psychological sub-scale: 6-weeks pre-baseline: number analyzed (Participants) | 8 | 10 | 18
  Psychological sub-scale: 6-weeks pre-baseline | NA (NA) — Data wasn't taken for the immediate intervention group at this timepoint. | 12.9 (3.98) | NA (NA) — Data wasn't taken for the immediate intervention group at this timepoint.
  Psychological sub-scale: Baseline | 11.63 (4.27) | 12.60 (3.91) | 12.16 (3.98)
  Psychological sub-scale: Imm. post-intervention | 11.88 (4.36) | 13.50 (4.25) | 12.79 (4.39)
  Psychological sub-scale:3 Months post-intervention | 11.75 (2.82) | 13.09 (2.77) | 12.53 (2.80)
  Psychological sub-scale:6 Months post-intervention | 11.00 (4.60) | 13.10 (3.53) | 12.21 (4.04)
  Psychological sub-scale:9 Months post-intervention: number analyzed (Participants) | 7 | 11 | 18
  Psychological sub-scale:9 Months post-intervention | 11.14 (4.06) | 12.45 (3.42) | 11.94 (3.62)
Statistical Analysis 1: Comparison: Immediate dk Leadership Intervention vs Delayed dk Leadership Intervention; Change in score in the immediate intervention group (after receiving the intervention for 6 weeks) compared to that of the delayed intervention group (after receiving no intervention for 6 weeks) for the physical component of the CIS; Test type: Superiority; p = 0.002, t-test, 2 sided; Cohen's d (effect size) = 1.792
Statistical Analysis 2: Comparison: Immediate dk Leadership Intervention vs Delayed dk Leadership Intervention; Change in score in the immediate intervention group (after receiving the intervention for 6 weeks) compared to that of the delayed intervention group (after receiving no intervention for 6 weeks) for the psychological component of the CIS; Test type: Superiority; p = 0.923, t-test, 2 sided; Cohen's d (effect size) = 0.047
Statistical Analysis 3: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of CIS (physical component) scores at baseline (pre-intervention) and immediately post-intervention; Test type: Superiority; p = 0.18, t-test, 2 sided; Cohen's d (effect size) = 0.60
Statistical Analysis 4: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of CIS (psychological component) scores at baseline (pre-intervention) and immediately post-intervention; Test type: Superiority; p = 0.388, t-test, 2 sided; Cohen's d (effect size) = 0.20
Statistical Analysis 5: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of CIS (physical component) scores at baseline (pre-intervention) and 3-months post-intervention; Test type: Superiority; p = 0.037, t-test, 2 sided; Cohen's d (effect size) = 0.52
Statistical Analysis 6: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of CIS (psychological component) scores at baseline (pre-intervention) and 3-months post-intervention; Test type: Superiority; p = 0.688, t-test, 2 sided; Cohen's d (effect size) = 0.09
Statistical Analysis 7: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of CIS (physical component) scores at baseline (pre-intervention) and 6-months post-intervention; Test type: Superiority; p = 0.038, t-test, 2 sided; Cohen's d (effect size) = 0.51
Statistical Analysis 8: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of CIS (psychological component) scores at baseline (pre-intervention) and 6-months post-intervention; Test type: Superiority; p = 0.956, t-test, 2 sided; Cohen's d (effect size) = 0.01
Statistical Analysis 9: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of CIS (physical component) scores at baseline (pre-intervention) and 9-months post-intervention; Test type: Superiority; p = 0.197, t-test, 2 sided; Cohen's d (effect size) = 0.32
Statistical Analysis 10: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of CIS (psychological component) scores at baseline (pre-intervention) and 9-months post-intervention; Test type: Superiority; p = 0.762, t-test, 2 sided; Cohen's d (effect size) = -0.07

3. Primary Outcome: Mean Change From Baseline in Social Connectedness Scores as Measured by the Social Connectedness Scale (SCS)
Description: Measured using the Social Connected Scale, a 20-item scale which measures belongingness - the degree to which people feel connected to others (internal consistency α = .92). Scores range from 20-120, with higher scores indicating greater social connectedness.
  Participants' scores at baseline will be compared with their scores post-intervention to detect changes in social connectedness. The change in scores over time will describe the general trajectory of social connectedness.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 8 | 11 | 19
score on a scale
  6-weeks pre-baseline: number analyzed (Participants) | 8 | 10 | 18
  6-weeks pre-baseline | NA (NA) — Data wasn't taken for the immediate intervention group at this timepoint. | 70.00 (10.10) | NA (NA) — Data wasn't taken for the immediate intervention group at this timepoint.
  Baseline (pre-intervention) | 74.00 (13.37) | 71.00 (15.60) | 72.26 (14.39)
  Immediately post-intervention | 75.75 (25.41) | 75.20 (14.60) | 75.42 (19.23)
  3-Months post-intervention | 82.88 (20.79) | 75.27 (8.46) | 78.47 (14.92)
  6-Months post-intervention | 84.38 (18.95) | 72.18 (12.36) | 77.32 (16.21)
  9-Months post-intervention: number analyzed (Participants) | 7 | 11 | 18
  9-Months post-intervention | 84.14 (14.81) | 73.26 (14.49) | 77.49 (15.19)
Statistical Analysis 1: Comparison: Immediate dk Leadership Intervention vs Delayed dk Leadership Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.834, t-test, 2 sided; Cohen's d (effect size) = 0.101
Statistical Analysis 2: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of SCS scores at baseline (pre-intervention) and immediately post-intervention; Test type: Superiority; p = 0.417, t-test, 2 sided; Cohen's d (effect size) = 0.19
Statistical Analysis 3: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of SCS scores at baseline (pre-intervention) and 3-months post-intervention; Test type: Superiority; p = 0.087, t-test, 2 sided; Cohen's d (effect size) = 0.42
Statistical Analysis 4: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of SCS scores at baseline (pre-intervention) and 6-months post-intervention; Test type: Superiority; p = 0.168, t-test, 2 sided; Cohen's d (effect size) = 0.33
Statistical Analysis 5: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of SCS scores at baseline (pre-intervention) and 9-months post-intervention; Test type: Superiority; p = 0.133, t-test, 2 sided; Cohen's d (effect size) = 0.37

4. Primary Outcome: Mean Change From Baseline in Self-esteem Scores as Measured by the Rosenberg Self-Esteem Scale (RSS)
Description: Assessed using the Rosenberg Self-Esteem Scale, a 10-item scale which measures of global self-worth (internal consistency α = .77 - .88). Scores range from 0-30. A score of <15 is categorized as low self-esteem, and 15-30 is categorized as normal self-esteem.
  Participants' scores at baseline will be compared with their scores post-intervention to detect changes in self-esteem. The change in scores over time will describe the general trajectory of self-esteem.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 8 | 11 | 19
score on a scale
  6-Weeks pre-baseline: number analyzed (Participants) | 8 | 10 | 18
  6-Weeks pre-baseline | NA (NA) — Data wasn't collected for the immediate intervention group at this timepoint. | 17.70 (4.91) | NA (NA) — Data wasn't collected for the immediate intervention group at this timepoint.
  Baseline (pre-intervention) | 16.66 (2.92) | 18.50 (6.09) | 17.70 (4.97)
  Immediately post-intervention | 22.00 (4.87) | 19.20 (7.31) | 20.37 (6.40)
  3-Months post-intervention | 21.00 (6.39) | 18.09 (5.11) | 19.32 (5.71)
  6-Months post-intervention | 24.75 (5.23) | 19.18 (6.88) | 21.53 (6.70)
  9-Months post-intervention: number analyzed (Participants) | 7 | 11 | 18
  9-Months post-intervention | 21.86 (4.98) | 19.00 (4.24) | 20.11 (4.63)
Statistical Analysis 1: Comparison: Immediate dk Leadership Intervention vs Delayed dk Leadership Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.026, t-test, 2 sided; Cohen's d (effect size) = 1.161
Statistical Analysis 2: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of RSS scores at baseline (pre-intervention) and immediately post-intervention; Test type: Superiority; p = 0.014, t-test, 2 sided; Cohen's d (effect size) = 0.62
Statistical Analysis 3: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of RSS scores at baseline (pre-intervention) and 3-months post-intervention; Test type: Superiority; p = 0.217, t-test, 2 sided; Cohen's d (effect size) = 0.29
Statistical Analysis 4: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of RSS scores at baseline (pre-intervention) and 6-months post-intervention; Test type: Superiority; p = 0.006, t-test, 2 sided; Cohen's d (effect size) = 0.71
Statistical Analysis 5: Comparison: Pooled Analysis of Immediate and Delayed Intervention Groups; Comparison of RSS scores at baseline (pre-intervention) and 9-months post-intervention; Test type: Superiority; p = 0.039, t-test, 2 sided; Cohen's d (effect size) = 0.53

5. Secondary Outcome: Change in Vocational Participation/Employment as Assessed by a Questionnaire From Baseline to 9-Months
Description: Acquirement of meaningful employment will be assessed. Participants will be prompted to answer questions about their current employment status, intensity of employment, and type of employment in the questionnaire. The change in the number of participants engaging in employment over time at the aggregate level will be assessed.
Time Frame: Assessed at baseline (immediately pre-intervention) and 9 months post-intervention
Population: 1 participant was lost to follow-up at the 9-month data collection period. Thus, the number of participants analyzed at 9-months is 18 rather than 19.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Analysis of Immediate and Delayed Intervention Groups: Data for the immediate and delayed intervention groups were pooled.
Arm/Group | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 19
Participants
  Baseline (pre-intervention): Full-time (>=30 hours/week) | 3
  Baseline (pre-intervention): Part-time (<30 hours/week) | 6
  Baseline (pre-intervention): Unemployed | 10
  9-Months post-intervention: number analyzed (Participants) | 18
  9-Months post-intervention: Full-time (>=30 hours/week) | 2
  9-Months post-intervention: Part-time (<30 hours/week) | 5
  9-Months post-intervention: Unemployed | 11

6. Secondary Outcome: Change in Academic Participation/Educational Attainment as Assessed by a Questionnaire From Baseline to 9-Months
Description: Participants will be prompted to answer questions about their current educational pursuit, and type of schooling or training program in a questionnaire. The change in the number of participants engaging in education over time on the aggregate will be assessed.
Time Frame: Assessed at baseline (immediately pre-intervention) and 9 months post-intervention
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 19
Participants
  Baseline (pre-intervention): Secondary education | 4
  Baseline (pre-intervention): Post-secondary education | 4
  Baseline (pre-intervention): Not pursuing education | 11
  9-Months post-intervention: number analyzed (Participants) | 18
  9-Months post-intervention: Secondary education | 1
  9-Months post-intervention: Post-secondary education | 7
  9-Months post-intervention: Not pursuing education | 10

7. Secondary Outcome: Number of Themes Related to Change in Career Awareness Informed by Focus Groups With Participants
Description: This outcome will describe the general trajectory of career awareness. Self-awareness, confidence, ability to articulate career goals, and understanding of how to achieve career goals will be assessed in focus groups. The questions posed during the focus groups will be guided by the evaluation objectives, but will be conversational and exploratory in nature with particular attention to identity capital, life-trajectories, and social inclusion. All will be conducted by the co-investigator at locations most convenient for the study participants, and will be audio recorded and transcribed verbatim. All focus groups will be analyzed together; the themes identified from the analysis will be presented as one data entry.
Time Frame: 60 - 90 minute focus groups at each of the following timepoints: immediately post-intervention, 3 months post-intervention, 6 months post-intervention, and 9 months post-intervention
Measure: Number; unit: Key themes identified
Arm/Group | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 19
Key themes identified
  Themes | 2
  Subthemes | 2

8. Secondary Outcome: Number of Themes Related to Change in Knowledge and Use of Soft Skills Informed by Focus Groups With Participants
Description: Acquirement of soft skills such as motivation, goal setting, self-discipline, and organization will be assessed in focus groups. The questions posed during the focus groups will be guided by the evaluation objectives, but will be conversational and exploratory in nature with particular attention to identity capital, life-trajectories, and social inclusion. All will be conducted by the co-investigator at locations most convenient for the study participants, and will be audio recorded and transcribed verbatim. All focus groups will be analyzed together; the themes identified from the analysis will be presented as one data entry.
Time Frame: as for outcome 7
Measure: Number; unit: Key themes identified
Arm/Group | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 19
Key themes identified
  Themes | 2
  Subthemes | 2

9. Secondary Outcome: Number of Themes Related to Participant Perspectives of Intervention Barriers and Facilitators, as Informed by Focus Groups With Participants
Description: In focus groups, youth will be prompted to discuss the strengths and drawbacks of conventional programs for youth transitioning out of homelessness. These evaluations will be compared to this intervention to determine what aspects of programs youth find most helpful, and which could be improved upon. The questions posed during the focus groups will be guided by the evaluation objectives, but will be conversational and exploratory in nature with particular attention to identity capital, life-trajectories, and social inclusion.All will be conducted by the co-investigator at locations most convenient for the study participants, and will be audio recorded and transcribed verbatim. All focus groups will be analyzed together; the themes identified from the analysis will be presented as one data entry.
Time Frame: as for outcome 7
Measure: Number; unit: Key themes identified
Arm/Group | Pooled Analysis of Immediate and Delayed Intervention Groups
Number analyzed (Participants) | 19
Key themes identified
  Themes | 2
  Subthemes | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time participants were enrolled to the end of the 9-month follow-up period. This was roughly 1 year for each participant.
Description: Our intervention was an identity-based intervention that proposed little risk to participants; thus no study-related adverse events were observed.
Arm/Group | Immediate dk Leadership Intervention | Delayed dk Leadership Intervention
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 0/8 | 0/11

LIMITATIONS AND CAVEATS:
A limitation is that the small sample size means the findings are unable to be generalized to young people in other contexts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT03772522/Prot_SAP_ICF_000.pdf